CLINICAL TRIAL: NCT02087631
Title: A Dose-finding, Safety and Tolerability Trial of Extended-release Quetiapine in Relapsing-remitting and Progressive Multiple Sclerosis
Brief Title: Safety and Tolerability of Quetiapine in Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Multiple Sclerosis Society of Canada (Other)
Responsible Party: Principal Investigator, Dr. Luanne Metz, Professor, University of Calgary
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QTPMS01
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; quetiapine; remyelination
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quetiapine (Experimental): Extended-release quetiapine fumarate up to 300mg once daily for 4 weeks
  Interventions: Drug: Extended-release quetiapine fumarate

INTERVENTIONS:
Drug: Extended-release quetiapine fumarate — Dosing schedule for RRMS: Group 1: Day 1-3:50 mg Day 4-6:100 mg Day 7-28:150 mg Day 29-30:100mg Day 31-32:50mg; Group 2: Day 1-2:50 mg Day 3-4:150 mg Day 5-6:200 mg Day 7-28:300 mg Day 29-30:250mg Day 31-32:200mg Day 33-34:150mg Day 35-36:100mg Day 37-38:50mg; Group 3: Day 1:50 mg Day 2:100 mg Day 3:200 mg Day 4-28:300 mg Day 29-30:250mg Day 31-32:200mg Day 33-34:150mg Day 35-36:100mg Day 37-38:50mg Dosing schedule for progressive MS: Group 1: Day 1-14: 50 mg Day 15-28: 100 mg Day 29-30: 50mg; Group 2: Day 1-5: 50 mg Day 6-10: 100 mg Day 11-15: 150 mg Day 16-28: 200 mg Day 29-30: 150mg Day 31-32: 100mg Day 33-34: 50mg; Group 3: Day 1-5: 50 mg Day 6-10: 100 mg Day 11-15: 200 mg Day 16-28: 300 mg Day 29-30: 250mg Day 31-32: 200mg Day 33-34: 150mg Day 35-36: 100mg Day 37-38: 50mg
  Other Names: Seroquel XR

SUMMARY:
Study Purpose:

The purpose of this clinical trial is to determine if extended-release quetiapine in a dose of 300 mg daily is tolerable to people with relapsing remitting and progressive MS. The investigators will also determine if the investigators can increase the dose up to 300 mg daily within 3 days in people with relapsing remitting MS and within 2 weeks in people with progressive MS. The investigators will determine if at least two thirds of study participants tolerate the drug well enough to continue it for 4 weeks. Tolerance will be determined separately for people with relapsing remitting and progressive MS. People with progressive MS may be less tolerant of side effects because of greater underlying brain injury from MS. Alternatively, people with progressive MS may gain more benefit from the improved sleep that usually occurs with use of quetiapine or they may be more willing to tolerate some side effects. This clinical trial will determine the maximally tolerated dose for future trials of this drug.

The number of participants in this study will depend on the tolerability at each dose tested. A maximum of 18 people with relapsing remitting MS and 18 people with primary or secondary progressive MS will be included.

Study Design:

The cohort expansion design (3+3) is used to determine toxicity-based dosing. This design is used in oncology phase I trials as it is guided by patient safety and minimizes the number of participants exposed to toxicity (Ivy et al. 2010). Maximum toxicity is defined as 33% or less. In this model, three patients will comprise the initial cohort. In the absence of DLT treatment may be escalated to the next higher dose in the next group of three patients. However, if one of three patients reaches DLT the cohort is expanded to six patients to verify that the toxicity rate has not exceeded or reached 33%. When the toxicity rate exceeds or reaches 33% in a cohort, this dose is deemed the maximum administered dose and a lower dose will be used in the next group of three patients. Patients with RRMS and progressive MS will be evaluated in separate groups using different dose schedules.

DETAILED DESCRIPTION:
Background:

Multiple sclerosis causes episodes of inflammation that injure or kill nerve cells and the cells that coat them with myelin. These episodes of inflammation may cause a relapse (attack) or the inflammation may only be detectable with brain MRI. Inflammatory episodes are the main feature of relapsing-remitting MS (RRMS). Most relapses can be prevented by current treatments for RRMS. This remains important because dead nerve cells cannot be replaced.

Fortunately, there are also repair processes that can rescue injured nerve and myelin cells. An important aspect of repair is regeneration of the myelin forming cells. If the myelin can be protected or even replaced the nerves have a better chance of survival. However if injured myelin is not repaired or replaced the nerve cell is not protected and will likely later also die; this may be the underlying process that causes the progression. The investigators obviously need therapies in MS that do more than just reduce the frequency of relapses and the silent episodes of inflammation. The investigators need treatments that help repair.

Quetiapine is a medication which has been shown to stimulate the myelin forming cells (called oligodendrocytes) to improve myelin repair in mice. It therefore may also improve myelin repair in people with MS. However, before testing the effects of quetiapine on myelin repair, the investigators must first determine if the medication is safe and if the dose is tolerated in people with MS in short-term treatment trials.

Quetiapine is currently approved in Canada to treat several psychiatric conditions including depression and psychosis. It has also been shown to be useful to treat anxiety and insomnia. Quetiapine is available as an extended release pill that can be taken once daily. Doses up to 800 mg per day may be used to treat some of these conditions but the investigators estimate that a dose of only 300 mg daily will be needed to stimulate myelin repair. It is not clear if the dose of 300 mg will be well tolerated by people with MS who may not need a medication to treat these conditions.

Visit schedule:

Screen period, baseline, week 1 [telephone], week 2 [telephone], week 3 [telephone], week 4, and week 8. Treatment with quetiapine XR will last for 4 weeks or until day 28. On day 29, the dose of quetiapine will be tapered by 50 mg every two days to avoid development of withdrawal syndrome and insomnia.

Treatment and Dose schedule:

Quetiapine XR dosing schedule for relapsing-remitting MS Group 1 Dose schedule Day 1-3: 50 mg Day 4-6: 100 mg Day 7-28: 150 mg Day 29-30: 100mg Day 31-32: 50mg Group 2 Dose schedule Day 1-2: 50 mg Day 3-4: 150 mg Day 5-6: 200 mg Day 7-28: 300 mg Day 29-30: 250mg Day 31-32: 200mg Day 33-34: 150mg Day 35-36: 100mg Day 37-38: 50mg Group 3 Dose Schedule Day 1: 50 mg Day 2: 100 mg Day 3: 200 mg Day 4-28: 300 mg Day 29-30: 250mg Day 31-32: 200mg Day 33-34: 150mg Day 35-36: 100mg Day 37-38: 50mg Quetiapine XR dosing schedule for progressive MS Group 1 Dose schedule Day 1-14: 50 mg Day 15-28: 100 mg Day 29-30: 50mg Group 2 Dose schedule Day 1-5: 50 mg Day 6-10: 100 mg Day 11-15: 150 mg Day 16-28: 200 mg Day 29-30: 150mg Day 31-32: 100mg Day 33-34: 50mg Group 3 Dose Schedule Day 1-5: 50 mg Day 6-10: 100 mg Day 11-15: 200 mg Day 16-28: 300 mg Day 29-30: 250mg Day 31-32: 200mg Day 33-34: 150mg Day 35-36: 100mg Day 37-38: 50mg

Measures:

1. Determination of dose-limiting toxicity Dose-limiting toxicity for any patient in this study is defined as early discontinuation of quetiapine XR due to an AE that is possibly, probably or definitely due to use of study drug. Patients who discontinue medication due to an AE will still be kept in the trial for safety assessment at weeks 4 and 8. Because of the small number of treated participants anyone who discontinues study drug for a reason or adverse event unrelated to use of the study drug will be excluded from the analysis and replaced. The dose-limiting toxicity will be determined for each group of patients: RRMS and progressive MS. The maximally tolerated dose and dose escalation schedule for future trials is the dose where fewer than 33% of participants reached dose-limiting toxicity. This will differ for each group of patients, RRMS and progressive MS.
2. Scales

   1. Functional Systems (FS) and Expanded Disability Status Scale (EDSS) A score based on a standardized neurological examination, observation of ambulation distance (up to 500 metres), and questions regarding bladder, bowel and sexual function.
   2. Extrapyramidal Symptom Rating Scale (ESRS) Neurological assessment of four extrapyramidal abnormalities: dystonia, dyskinesia, parkinsonism, akathisia, as well as subjective extrapyramidal symptoms
   3. 9-hole Peg Test (9-HPT) Timed test of arm/hand function
   4. Timed 25-Foot Walk (T25-FW) Timed test of ambulation
   5. Symbol Digit Modalities Test (SDMT) Timed test of cognitive processing speed and working memory
   6. Epworth Sleepiness Scale (ESS) 8 self-report items measuring sleepiness
   7. Modified Fatigue Impact Scale (MFIS) 21 self-report items measuring fatigue
   8. Athens Insomnia Scale (AIS) 8 self-report items measuring insomnia
   9. Center for Epidemiologic Studies Depression Scale (CES-D) 20 self-report items measuring depression

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Sexually active men and women of child-bearing potential, defined as those who are not postmenopausal (24 consecutive months) or permanently sterilised, must agree to use adequate contraception. Adequate contraception is defined as methods of birth control which result in a low failure rate [i.e. less than 1% per year] when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), barrier contraceptives, sexual abstinence or vasectomised partner. Adequate contraception is required during quetiapine treatment and for one month after stopping treatment.
* MS defined according to the McDonald criteria (2010; Polman et al. 2011)
* Progressive MS (primary progressive course, secondary progressive course, or progressive relapsing course) course according to Lublin and Reingold (1996).

NOTE: No longer recruiting RRMS patients

* Patients currently on glatiramer acetate, interferon-beta, fingolimod (treatment longer than 3 months), or dimethyl fumarate as well as those on no treatment.
* Written informed consent

Exclusion Criteria:

Patients are to be excluded from enrolment if they display any of the following (current treatment reflects use at the time of screening and 14 days before screening):

* Clinically significant depression, renal, hepatic, cardiovascular, respiratory, metabolic, ophthalmologic, cerebrovascular, or other serious physical disease
* Inability to perform the 9 hole peg test and the oral SDMT at baseline
* Diagnosis of dementia, diabetes, or cataracts
* History of seizures, tardive dyskinesia, or symptomatic hypotension.
* Clinically significant gastrointestinal or endocrine disorder, such as pancreatitis, gastrointestinal obstruction, and hypothyroidism
* Poorly managed constipation, defined as a bowel routine that does not result in a bowel movement at least every other day.
* The presence of any circumstances that may increase the risk of occurrence of torsade de pointes and/or sudden death including (1) a history of cardiac arrhythmias such as bradycardia; (2) hypokalemia or hypomagnesaemia; (3) concomitant use of other drugs that prolong the QTc interval; (4) prolonged QTc at screening; and (5) presence of congenital prolongation of the QT interval
* Body Mass Index > 30 (obesity)
* Clinically significant abnormal laboratory values, electrocardiogram, or vital signs at screening or any elevation of fasting glucose
* Pregnant or breastfeeding women
* Current treatment with natalizumab
* Current treatment with immunosuppressive medications other than: steroids for relapses and the MS disease-modifying therapies mentioned in the inclusion criteria. Initiation of fingolimod within the previous 3 months
* Substances that are not permitted include current treatment with: potent CYP3A4 inhibitors (e.g. ketoconazole, ritonavir) or potent CYP3A4 inducers (e.g. phenytoin, rifampin, St. John's Wort), pro- or anti-dopaminergic medications, or medications that produce clinically significant alterations of QTc interval.
* Previous or current treatment with quetiapine or any other antipsychotic
* Known hypersensitivity to any of the ingredients in quetiapine including lactose
* Inability to swallow pills without chewing or crushing
* Use, within the previous three months, of any experimental MS treatment
* Any other condition or situation that in the opinion of the investigator would either put the patient at risk of worsening health if enrolled in the trial or would prevent completion of the trial
* Concurrent participation in any therapeutic clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | 4 weeks
  The primary outcome is the occurrence of dose-limiting toxicity (DLT). Dose-limiting toxicity for any patient in this study is defined as early discontinuation of quetiapine XR due to an adverse event (AE) that is possibly, probably or definitely due to use of study drug. Patients who discontinue medication due to an AE will still be kept in the trial for safety assessment at weeks 4 and 8. Because of the small number of treated participants anyone who discontinues study drug for a reason or adverse event unrelated to use of the study drug will be excluded from the analysis and replaced. The dose-limiting toxicity will be determined for each group of patients: RRMS and progressive MS by the week 4 visit.

SECONDARY OUTCOMES:
Adverse events | 4 weeks
  Secondary objectives are to determine treatment safety and tolerance. This will be determined by adverse event reporting; by measuring the impact of treatment on sleep, fatigue, and depression using validated patient report scales; by determining the occurrence of extrapyramidal function by using the extrapyramidal symptom rating scale; and by measuring the impact on cognition by means of the symbol digit modality test.

CONTACTS AND LOCATIONS:
Overall Officials: Luanne M Metz, MD,FRCPC, Principal Investigator — University of Calgary
Locations (1):
- MS Clinic, Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
consent was not obtained from subjects so data can not be shared

REFERENCES:
- [Background] Zhornitsky S, Wee Yong V, Koch MW, Mackie A, Potvin S, Patten SB, Metz LM. Quetiapine fumarate for the treatment of multiple sclerosis: focus on myelin repair. CNS Neurosci Ther. 2013 Oct;19(10):737-44. doi: 10.1111/cns.12154. Epub 2013 Jul 22. PMID 23870612